CLINICAL TRIAL: NCT06493162
Title: Comparison of Flow Controlled Ventilation and Volume Controlled Ventilation in Microscopic Laryngeal Surgeries, a Randomized Controlled Trial
Brief Title: Comparison of Flow Controlled Ventilation and Volume Controlled Ventilation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Hadi Ufuk Yörükoğlu, Principal investigator, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: KAEK/05.bI.07
Record Dates: First submitted 2024-06-29; First posted 2024-07-09 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Vocal Cord Disease; Vocal Cord Cyst
Keywords: Microscopic Laryngeal Surgery; Flow Controlled Ventilation; Volume Controlled Ventilation
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FCV Group (Active Comparator): Patients who will be ventilated with flow controlled ventilation following the intubation
  Interventions: Procedure: Intubation; Device: Flow Controlled Ventilation
- VCV Group (Active Comparator): Patients who will be ventilated with volume controlled ventilation following the intubation
  Interventions: Procedure: Intubation; Device: Volume Controlled Ventilation

INTERVENTIONS:
Procedure: Intubation — Patients will be intubated with 5mm sized endotracheal tube for microscopic laryngeal surgery
Device: Flow Controlled Ventilation — Patients in FCV group will be ventilated with flow controlled ventilation mode
  Arms: FCV Group
Device: Volume Controlled Ventilation — Patients in VCV group will be ventilated with volume controlled ventilation mode
  Arms: VCV Group

SUMMARY:
Flow-Controlled Ventilation is designed to ventilate the patient with constant flows during both inspiration and expiration. During inspiration, the pressure rises linearly from a set positive end-expiratory pressure (PEEP) to a set positive inspiratory pressure (PIP), and then falls linearly from PIP to end-expiratory pressure (EEP) during expiration. There are no flow interruptions during the Flow-Controlled Ventilation cycle, and the rate of change of pressure and volume in the lungs is equal, allowing for higher tidal volumes at lower pressures. The user sets the inspiratory flow rate and the ratio of inspiratory to expiratory time, providing full control over the ventilation cycle. However, this results in two unusual features: During inspiration, the ventilator creates positive pressure to direct gas into the patient's lungs through the endotracheal tube (ETT). When the intratracheal pressure (airway pressure) reaches the set PIP value, the ventilator switches from inspiration to expiration. By reversing the flow, it utilizes the Bernoulli effect to create negative pressure, facilitating expiration. Despite the presence of negative pressure on the ventilator side, the pressure in the patient's airway remains positive at all times.

Volume-controlled ventilation is a mode that is volume-controlled, time-cycled, time-triggered, and pressure-limited. In volume-controlled ventilation, high pressures are sometimes necessary to reach the target tidal volume. This can lead to barotrauma, atelectrauma, and volutrauma in the lungs. Therefore, to avoid high pressures, low tidal volume ventilation is preferred.

For Microscopic Laryngeal Surgeries, patients are intubated with a small sized endotracheal tube which results with higher pressures. We think that flow controlled ventilation will improve the ventilation during the surgery with lower pressures.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo elective microscopic laser surgery
* ASA status I and II

Exclusion Criteria:

* Surgery time more than 2 hours
* Patients with difficult intubation
* Patients with chronic lung diseases
* BMI > 25

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
PIP | 10 minutes interval after the intubation during the surgery
  Peak inspiratory pressure
RR | 10 minutes interval after the intubation during the surgery
  Respiratory rate
TV | 10 minutes interval after the intubation during the surgery
  Tidal volume
Compliance (Cdyn) | 10 minutes interval after the intubation during the surgery
  Dynamic compliance (ventilator calculates: Cdyn = tidal volume/(PIP - PEEP)
Resistance | 10 minutes interval after the intubation during the surgery
  Resistance (ventilator calculates: dividing the [peak pressure minus the plateau pressure] by the flowrate in litres per second)

SECONDARY OUTCOMES:
HR | 10 minutes interval after the intubation during the surgery
  Heart rate
MP | 10 minutes interval after the intubation during the surgery
  Mean blood pressure
SpO2 | 10 minutes interval after the intubation during the surgery
  Oxygen saturation

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No